CLINICAL TRIAL: NCT03660540
Title: Improving Preoperative Screening and Postoperative Nutrition in Orthopedic Sarcoma and Spine Patients: Pilot Study
Brief Title: Spine and Tumor Screening and Supplementation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No enrollment
Sponsor: University of Iowa (Other)
Collaborators: Orthopaedic Trauma Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 201805970
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Spinal Injuries; Sarcoma; Nutritional Deficiency
MeSH Terms: conditions — Spinal Injuries; Sarcoma; Malnutrition

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutritional supplement group (Experimental): Subjects in this group will be asked to consume the nutritional supplement on a daily basis, in addition to standard nutrition. Subjects will have pain medication and postoperative therapies per standard of care.
  Interventions: Dietary Supplement: Juven
- Standard nutrition group (No Intervention): Subjects in this group will have standard nutrition provided per dietitian recommendation. Subjects will have pain medication and postoperative therapies per standard of care.

INTERVENTIONS:
Dietary Supplement: Juven — Nutritional supplement (Juven) will be consumed daily per manufacturer recommendations.
  Arms: Nutritional supplement group

SUMMARY:
This project aims to evaluate an implementable screening tool and nutritional interventions that will lead to improved quality and patient safety. The aims of this pilot study are twofold:

Purpose 1: assess the prognostic value of malnutrition and sarcopenia for identifying patients at increased risk of adverse postoperative outcomes following elective or semi-elective orthopedic procedures.

Purpose 2: assess the clinical benefit of postoperative oral supplementation with a commercially-available nutritional supplement that includes conditionally-essential branched chain amino acids.

DETAILED DESCRIPTION:
All patients will be treated according to standard of care for their orthopedic injuries, including standard nutritional support in the preoperative period. Patients admitted to our academic Level I trauma center with spinal fractures and sarcoma requiring limb reconstruction will be approached for consent to participate in this study. Consented patients will be prospectively enrolled at the time of admission. We will obtain relevant patient medical history, standard preoperative labs, radiographic imaging, and nutritional assessment at the time of admission. Patients will be assessed for the presence of sarcopenia utilizing ultrasound measures of skeletal muscle as previously described.

All patients will be evaluated by a clinical dietitian or dietetic assistant for nutritional assessment as part of the standard of care. In addition to screening for sarcopenia and malnutrition, we will assess the clinical benefit of oral nutritional supplementation with essential branched-chain amino acids in a population of trauma patients. Patients providing written informed consent will be enrolled in a prospective RCT to assess nutritional supplementation with conditionally essential branched-chain amino acids. Patients will be randomly assigned to receive standard nutritional support or standard nutrition plus oral supplementation with a commercially available nutritional supplement containing essential branched chain amino acids (Juven, Abbot Nutrition). Similar combinations of essential amino acids have previously demonstrated protective effects against skeletal muscle wasting and medical complications in immobilized critically ill patients. Patients will be prospectively followed for 12 months from the time of admission to assess clinical outcomes. Our primary outcome measures include skeletal muscle mass changes, wound healing complications,

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Indicated for spinal or orthopedic oncology surgery

Exclusion Criteria:

* Unable to provide written consent
* Unable to comply with postoperative treatment recommendations
* Do not plan to follow up at the facility where surgery occurred
* Food allergy to ingredients in dietary supplement
* Intolerance to oral diet including phenylketonuria
* Pregnant women
* Individuals with dementia
* Vulnerable populations (minors, prisoners)
* Individuals lacking decision making capacity

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Body composition | One year
  Change in muscle mass

SECONDARY OUTCOMES:
Hand grip strength | One year
  Change in hand grip strength as measured by hand held dynamometer
Post-operative complications | One year
  Medical and surgical complications following operative fracture fixation, validated patient

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Hendrickson, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No